CLINICAL TRIAL: NCT07231263
Title: The Effect of Human Papillomavirus Education Provided to Women on Their Level of Knowledge Regarding Human Papillomavirus
Brief Title: Effect of HPV Education on Women's Knowledge
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Fatma Keskin Töre, ASSOCIATE PROFESSOR, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025/23/04
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Human Papillomavirus (HPV); Awareness and Knowledge Level
Keywords: Human papillomavirus (HPV); HPV education; Women's health;

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV Awareness Education Group (Experimental)
  Interventions: Other: HPV Awareness Education Group
- Control Group (No Intervention)

INTERVENTIONS:
Other: HPV Awareness Education Group — Women who agree to participate in the training will receive a total of two hours of HPV awareness training in two sessions on the predetermined training date. The HPV awareness training will be delivered using a PowerPoint presentation, and at the end of the training, a brochure created in line with the literature will be distributed to the participating women to ensure retention. The brochure will be prepared by the researcher based on current literature sources. Expert opinions will be sought from specialists in the field of obstetrics and gynecology nursing regarding the training content, and revisions will be made if necessary. The training content will include the definition of HPV, risk factors, etiology, screening, HPV vaccination, transmission and prevention methods, and treatment. The training topics will be prepared by the faculty members responsible for the research in accordance with the literature.
  Arms: HPV Awareness Education Group

SUMMARY:
This interventional study aims to evaluate the effectiveness of an educational program on women's knowledge of Human Papillomavirus (HPV), HPV vaccination, and screening. HPV is a major public health concern worldwide and a leading cause of cervical cancer. Although cervical cancer is preventable through vaccination and early screening, HPV awareness among women remains limited in Türkiye. Educational interventions are therefore essential to improve knowledge and promote preventive health behaviors.

The study population consists of 110 women attending courses at the Suzan and Abdulhakim Bilgili Public Education Center in Onikişubat, Kahramanmaraş, Türkiye, between August 2025 and December 2025. No formal sample size calculation was performed. Instead, 80 women who met the inclusion criteria and voluntarily agreed to participate were included in the study.

Participants were randomly assigned to either the intervention group (education) or the control group (no education). The HPV education program is delivered in two 1-hour sessions using PowerPoint presentations and informational brochures developed from current literature and reviewed by experts in women's health nursing.

Data are collected before and after the educational sessions using a Personal Information Form and the HPV Knowledge Scale (HPV-KS), which measures participants' knowledge about HPV infection, vaccination, and screening. Statistical analyses will be conducted using SPSS 22.0, with descriptive statistics and inferential tests (paired-sample t-test, independent-sample t-test, repeated-measures ANOVA, and non-parametric equivalents) applied as appropriate. A p-value < 0.05 will be considered statistically significant.

It is hypothesized that women receiving HPV education will demonstrate significantly higher post-intervention knowledge scores compared to those in the control group.

DETAILED DESCRIPTION:
Human papillomavirus (HPV) is a highly contagious virus that is recognized as a major public health problem both nationally and internationally due to its association with cervical cancer. Cervical cancer is a type of cancer within the category of gynecological cancers that can be detected early through screening programs, thereby preventing its progression. It ranks fourth among the most common cancers in women and remains a leading cause of cancer-related deaths. Globally, in 2020, there were 604,000 new cervical cancer cases and 342,000 deaths caused by cervical cancer. The World Health Organization recommends the inclusion of HPV vaccines in national immunization programs. While HPV vaccination rates are high in developed countries, there are delays in vaccine access in underdeveloped and developing countries . In Türkiye, HPV vaccination has not yet been incorporated into the national immunization program.

Cervical cancer remains one of the leading health concerns worldwide in terms of mortality and morbidity rates. The high incidence, insufficient HPV screening, and low awareness of HPV indicate the widespread presence of HPV infection . Increasing public awareness, preventing disease occurrence, and implementing protective planning and educational interventions are of great importance. One of the key strategies for addressing cervical cancer is to promote HPV screening .

In Türkiye, several studies have been conducted to assess the level of knowledge about HPV and its vaccine among healthcare personnel and students in health-related fields. The results of these studies have shown that participants' knowledge about HPV is not at the desired level . These studies revealed deficiencies in fundamental areas such as HPV-related infections, vaccination methods, and the effectiveness and importance of the vaccine. Such knowledge gaps may limit healthcare professionals' ability to provide effective health services and raise public awareness regarding HPV. Similarly, studies evaluating women's knowledge, attitudes, and behaviors about HPV and its vaccine have generally shown that women's knowledge of HPV is low

Therefore, HPV education is considered highly important. Educational programs can help participants make informed decisions and protect their sexual health. The findings obtained from such programs may guide the implementation of similar initiatives for larger communities and increase awareness about HPV. These kinds of studies play a crucial role in designing preventive measures and awareness-raising programs for public health, while also contributing to the limited existing literature. Accordingly, this study aims to examine the effect of HPV education provided to women on their level of knowledge regarding human papillomavirus.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Agreeing to participate in the study,
* Not experiencing communication difficulties,
* Female students who complete the data collection form in full will be included in the study.

Exclusion Criteria:

* Previously tested positive for HPV
* History of cervical cancer
* Unreachable
* Not attending public education during the training period
* Female students who did not complete the data collection form will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-11-14 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
HPV knowledge level measured by the Human Papillomavirus Knowledge Scale (HPV-BÖ) | Baseline (pre-test) and immediately after the education session (post-test)
  his outcome will assess changes in participants' knowledge about HPV, HPV vaccination, HPV screening tests, and the national vaccination program using the HPV Knowledge Scale adapted to Turkish women. The scale consists of 33 items scored as 0-33, with higher scores indicating higher knowledge.

SECONDARY OUTCOMES:
General HPV knowledge measured by the HPV Knowledge Scale (HPV-BÖ) - Subscale 1 | Baseline and immediately after the intervention
  Evaluates participants' general knowledge about HPV infection using the related subscale of the HPV Knowledge Scale
Knowledge of HPV screening tests measured by the HPV Knowledge Scale (HPV-BÖ) - Subscale 2 | Baseline and immediately after the intervention
  Assesses changes in knowledge related to HPV screening tests
Knowledge of HPV vaccination measured by the HPV Knowledge Scale (HPV-BÖ) - Subscale 3 | Baseline and immediately after the intervention
  Assesses participants' knowledge about HPV vaccination and recommendations.
Knowledge of the national HPV vaccination program measured by the HPV Knowledge Scale (HPV-BÖ) - Subscale 4 | Baseline and immediately after the intervention
  Evaluates changes in awareness regarding the national HPV vaccination program.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. World Health Organization-WHO. Updates recommendations on HpV vacci- nation schedule